CLINICAL TRIAL: NCT02616497
Title: Comparison of Triflusal With Aspirin in the Secondary Prevention of Atherothrombotic Events
Brief Title: ASpirin vs Triflusal for Event Reduction In Atherothrombosis Secondary Prevention (ASTERIAS)
Acronym: ASTERIAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Alexandros Tselepis, Professor of Biochemistry and Clinical Chemistry, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Asp-Trifl-1
Record Dates: First submitted 2015-11-20; First posted 2015-11-30 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Atherothrombosis
Keywords: aspirin; triflusal; antiplatelet drugs; atherothrombosis; secondary prevention; bleeding
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Aspirin; triflusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Active Comparator): 100mg/day
  Interventions: Drug: Aspirin
- Triflusal (Active Comparator): 300mg twice or 600mg once daily
  Interventions: Drug: Triflusal

INTERVENTIONS:
Drug: Aspirin — COX-1 inhibitor
  Other Names: Salospir
  Arms: Aspirin
Drug: Triflusal — COX-1 inhibitor
  Other Names: Aflen
  Arms: Triflusal

SUMMARY:
Investigation of the efficacy and safety of triflusal in comparison with aspirin in patients with stable coronary artery disease (CAD) and in those with a history of an acute non-cardioembolic ischemic stroke.

DETAILED DESCRIPTION:
Triflusal, 2-(acetyloxy)-4-(trifluoromethyl) benzoic acid, is an antiplatelet agent with a chemical structure similar to aspirin, but with a different pharmacokinetic and pharmacodynamic profile. The drug is administered orally and its bioavailability ranges from 83% to 100%. It binds almost entirely (99%) to plasma proteins and crosses readily organic barriers. Triflusal is deacetylated in the liver, forming its main metabolite 2-hydroxy-4-trifluoromethyl benzoic acid (HTB). In contrast to the inactive aspirin metabolite salicylic acid, HTB exhibits antiplatelet activity and has a long plasma half-life of approximately 40h. Triflusal irreversibly inhibits COX-1 and reduces TxA2 production, but to a lesser extent compared with aspirin. It inhibits COX-1 and AA metabolism selectively in platelets, preserving PGI2 synthesis in vascular endothelial cells 1. Except of platelet COX-1 triflusal and in particular HTB inhibit phosphodiesterase, the enzyme that degrades the cyclic nucleotides, cyclic adenosine monophosphate (c-AMP) and cyclic guanosine monophosphate (c-GMP), both of which inhibit platelet function.

Triflusal has similar to aspirin efficacy for the secondary prevention of vascular events in patients with acute myocardial infarction (MI) and stroke, while it reduces the incidence of intracranial and gastrointestinal haemorrhage compared with aspirin. It should be noted that triflusal is well tolerated in patients with aspirin-induced asthma.

Aspirin (acetyl salicylic acid) remains for over 50 years the cornerstone of antiplatelet therapy due to its proven clinical benefit and very good cost effectiveness profile. Aspirin selectively and irreversibly acetylates the hydroxyl group of a single serine residue at position 529 within the polypeptide chain of PGH synthase-1. Thus aspirin inhibits the COX-1 activity but it does not affect the hydroperoxidase activity PGH synthase-1. By blocking COX-1, the production of TXA2 is reduced, leading to reduced platelet aggregation. Aspirin improves clinical outcome in all cardiovascular syndromes in primary and secondary prevention, including acute events. In high-risk patients, aspirin substantially reduces the risk of vascular death by ~15% and non-fatal vascular events by ~30% as it reported by a meta-analysis of over 100 large-scale randomized trials. Several studies the last years have suggested that a proportion of patients (5 to 65%) exhibit a hyporesponsiveness (resistance) to aspirin treatment which could be associated with recurrent ischemic events. Aspirin resistance may result from several causes, such as low compliance, interference with non-steroid anti-inflammatory drugs (NSAIDS) and protein glycation occurring in type 2 diabetes mellitus. Increased platelet turnover observed in various diseases such as ACS, peripheral arterial disease and diabetic angiopathy associated with faster re-appearance of newly formed, non aspirinated platelets, may also account for aspirin resistance.

Although triflusal is chemically related to aspirin and has similar effectiveness, it appears to have a better tolerability profile than aspirin. Results from large-scale clinical trials and a meta-analysis suggest that its use may be preferable to that of aspirin, in several clinical settings where antiplatelet therapy is indicated. Furthermore, in selected populations, such as in geriatric patients, because of an increased risk of bleeding complications, in patients suffering from asthma, chronic sinusitis and nasal polyps, or in cases of aspirin resistance, triflusal may be a choice worth considering. Furthermore, when combination antiplatelet-fibrinolytic or antiplatelet-anticoagulant therapy is needed, clinical data support triflusal use based on its efficacy and better safety than aspirin. Unlike aspirin, triflusal, also, less likely affect the efficacy of antihypertensive drugs, especially angiotensin converting enzyme inhibitors. The aim of the present trial is to investigate the efficacy and safety of triflusal in comparison with aspirin in patients with stable coronary artery disease (CAD) and in those with a history of an acute non-cardioembolic ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a stable coronary artery disease (CAD)
* Patients with a history of non-cardioembolic ischemic stroke.

Exclusion Criteria:

* Hypersensitivity reaction or contraindication to triflusal or aspirin
* Active bleeding or history of severe bleeding (peptic ulcer, trauma or intracranial hemorrhage)
* Blood coagulation disorders
* Uncontrolled severe hypertension
* Pregnancy or breastfeeding
* Liver disease (alanine or aspartate aminotransferase more than 3 times the upper normal limit)
* Malignancy that may potentially increase the risk of hemorrhage
* Drug or alcohol abuse
* HIV infection
* Chronic disorders requiring long-term treatment with systemic nonsteroidal anti-inflammatory drugs (NSAIDs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Composite of death from vascular causes, myocardial infarction (MI), or stroke (ischaemic or haemorrhagic) during the twelve month treatment period | 12 months
  Number of participants who suffer from the primary efficacy end point which is the composite of death from vascular causes, myocardial infarction(MI), or stroke during the twelve month treatment period
Rate of bleeding events as defined by Bleeding Academic Research Consortium (BARC) criteria during the twelve month treatment period | 12 months
  Number of participants who suffer from the rate of bleeding events as defined by Bleeding Academic Research Consortium (BARC) criteria during the twelve month treatment period

SECONDARY OUTCOMES:
Composite of death from any cause, MI, or stroke during the twelve month treatment period | 12 months
  Number of participants who suffer from the secondary efficacy end point which is the composite of death from any cause, MI, or stroke during the twelve month treatment period
Hypersensitivity or intolerance to study drugs during the twelve month treatment period | 12 months
  Number of participants who suffer from the secondary safety end points which are hypersensitivity or intolerance to study drugs during the twelve month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Tselepis, MD, Principal Investigator — Atherothrombosis Research Centre
Locations (1):
- Atherothrombosis Research Centre / Laboratory of Biochemistry, University of Ioannina, Ioannina, Greece

REFERENCES:
- [Background] Di Minno G. Aspirin resistance and platelet turnover: a 25-year old issue. Nutr Metab Cardiovasc Dis. 2011 Aug;21(8):542-5. doi: 10.1016/j.numecd.2011.04.002. Epub 2011 Jul 13. PMID 21745731
- [Background] Feher G, Feher A, Pusch G, Lupkovics G, Szapary L, Papp E. The genetics of antiplatelet drug resistance. Clin Genet. 2009 Jan;75(1):1-18. doi: 10.1111/j.1399-0004.2008.01105.x. Epub 2008 Nov 29. PMID 19067731
- [Background] Anninos H, Andrikopoulos G, Pastromas S, Sakellariou D, Theodorakis G, Vardas P. Triflusal: an old drug in modern antiplatelet therapy. Review of its action, use, safety and effectiveness. Hellenic J Cardiol. 2009 May-Jun;50(3):199-207. No abstract available. PMID 19465361
- [Background] Valle M, Barbanoj MJ, Donner A, Izquierdo I, Herranz U, Klein N, Eichler HG, Muller M, Brunner M. Access of HTB, main metabolite of triflusal, to cerebrospinal fluid in healthy volunteers. Eur J Clin Pharmacol. 2005 Apr;61(2):103-11. doi: 10.1007/s00228-004-0887-0. Epub 2005 Feb 12. PMID 15711832
- [Background] Antonijoan RM, Gich I, Azaro A, Sainz S, Balanzo J, Izquierdo I, Borja J, Donado E, Blanch I, Barbanoj MJ. Gastrointestinal safety of triflusal solution in healthy volunteers: a proof of concept endoscopic study. Eur J Clin Pharmacol. 2011 Jul;67(7):663-9. doi: 10.1007/s00228-011-1004-9. Epub 2011 Feb 16. PMID 21327422
- [Background] Michelson AD. Antiplatelet therapies for the treatment of cardiovascular disease. Nat Rev Drug Discov. 2010 Feb;9(2):154-69. doi: 10.1038/nrd2957. PMID 20118963
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Krasopoulos G, Brister SJ, Beattie WS, Buchanan MR. Aspirin "resistance" and risk of cardiovascular morbidity: systematic review and meta-analysis. BMJ. 2008 Jan 26;336(7637):195-8. doi: 10.1136/bmj.39430.529549.BE. Epub 2008 Jan 17. PMID 18202034
- [Background] Snoep JD, Hovens MM, Eikenboom JC, van der Bom JG, Huisman MV. Association of laboratory-defined aspirin resistance with a higher risk of recurrent cardiovascular events: a systematic review and meta-analysis. Arch Intern Med. 2007 Aug 13-27;167(15):1593-9. doi: 10.1001/archinte.167.15.1593. PMID 17698681
- [Background] Undas A, Siudak Z, Topor-Madry R, Lesniak M, Tracz W. Simvastatin administration reduces thromboxane production in subjects taking aspirin: links between aspirin resistance and thrombin generation. Int J Cardiol. 2012 Jan 12;154(1):59-64. doi: 10.1016/j.ijcard.2010.09.093. Epub 2010 Oct 29. PMID 21035882
- [Background] Acikel S, Yildirir A, Aydinalp A, Demirtas K, Bal U, Kaynar G, Ozin B, Karakayali H, Muderrisoglu H, Haberal M. Incidence of aspirin resistance and its relationship with cardiovascular risk factors and graft function in renal transplant recipients. Transplant Proc. 2008 Dec;40(10):3485-8. doi: 10.1016/j.transproceed.2008.06.108. PMID 19100419
- [Background] Simon DI, Jozic J. Drug-eluting stents and antiplatelet resistance. Am J Cardiol. 2008 Nov 3;102(9 Suppl):29J-37J. doi: 10.1016/j.amjcard.2008.09.007. PMID 18928790
- [Background] Papathanasiou A, Goudevenos J, Tselepis AD. Resistance to aspirin and clopidogrel: possible mechanisms, laboratory investigation, and clinical significance. Hellenic J Cardiol. 2007 Nov-Dec;48(6):352-63. No abstract available. PMID 18196658
- [Background] Kalantzi KI, Tsoumani ME, Goudevenos IA, Tselepis AD. Pharmacodynamic properties of antiplatelet agents: current knowledge and future perspectives. Expert Rev Clin Pharmacol. 2012 May;5(3):319-36. doi: 10.1586/ecp.12.19. PMID 22697594
- [Background] Murdoch D, Plosker GL. Triflusal: a review of its use in cerebral infarction and myocardial infarction, and as thromboprophylaxis in atrial fibrillation. Drugs. 2006;66(5):671-92. doi: 10.2165/00003495-200666050-00009. PMID 16620146
- [Background] Matias-Guiu J, Ferro JM, Alvarez-Sabin J, Torres F, Jimenez MD, Lago A, Melo T; TACIP Investigators. Comparison of triflusal and aspirin for prevention of vascular events in patients after cerebral infarction: the TACIP Study: a randomized, double-blind, multicenter trial. Stroke. 2003 Apr;34(4):840-8. doi: 10.1161/01.STR.0000063141.24491.50. Epub 2003 Mar 20. PMID 12649515
- [Background] Culebras A, Rotta-Escalante R, Vila J, Dominguez R, Abiusi G, Famulari A, Rey R, Bauso-Tosselli L, Gori H, Ferrari J, Reich E; TAPIRSS investigators. Triflusal vs aspirin for prevention of cerebral infarction: a randomized stroke study. Neurology. 2004 Apr 13;62(7):1073-80. doi: 10.1212/01.wnl.0000113757.34662.aa. PMID 15079004
- [Background] Cruz-Fernandez JM, Lopez-Bescos L, Garcia-Dorado D, Lopez Garcia-Aranda V, Cabades A, Martin-Jadraque L, Velasco JA, Castro-Beiras A, Torres F, Marfil F, Navarro E. Randomized comparative trial of triflusal and aspirin following acute myocardial infarction. Eur Heart J. 2000 Mar;21(6):457-65. doi: 10.1053/euhj.1999.1874. PMID 10681486
- [Background] Costa J, Ferro JM, Matias-Guiu J, Alvarez-Sabin J, Torres F. Triflusal for preventing serious vascular events in people at high risk. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD004296. doi: 10.1002/14651858.CD004296.pub2. PMID 16034926
- [Background] Perez-Gomez F, Alegria E, Berjon J, Iriarte JA, Zumalde J, Salvador A, Mataix L; NASPEAF Investigators. Comparative effects of antiplatelet, anticoagulant, or combined therapy in patients with valvular and nonvalvular atrial fibrillation: a randomized multicenter study. J Am Coll Cardiol. 2004 Oct 19;44(8):1557-66. doi: 10.1016/j.jacc.2004.05.084. PMID 15489085
- [Derived] Kalantzi KI, Ntalas IV, Chantzichristos VG, Tsoumani ME, Adamopoulos D, Asimakopoulos C, Bourdakis A, Darmanis P, Dimitriadou A, Gkiokas S, Ipeirotis K, Kitikidou K, Klonaris I, Kostaki A, Logothetis D, Mainas K, Mais T, Maragiannis A, Martiadou K, Mavronasos K, Michelongonas I, Mitropoulos D, Papadimitriou G, Papadopoulos A, Papaioakeim M, Sofillas K, Stabola S, Stefanakis E, Stergiou D, Thoma M, Zenetos A, Zisekas S, Goudevenos JA, Panagiotakos DB, Tselepis AD. Comparison of Triflusal with Aspirin in the Secondary Prevention of Atherothrombotic Events; Alpha Randomised Clinical Trial. Curr Vasc Pharmacol. 2019;17(6):635-643. doi: 10.2174/1570161116666180605090520. PMID 29866011